CLINICAL TRIAL: NCT05169411
Title: Preserving Kidney Function in Children With Chronic Kidney Disease (PRESERVE)
Brief Title: Preserving Kidney Function in Children With Chronic Kidney Disease
Acronym: PRESERVE
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Children's Hospital Medical Center, Cincinnati (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Nationwide Children's Hospital (Other); Seattle Children's Hospital (Other); Stanford University (Other); University of Colorado, Denver (Other); Duke University (Other); University of North Carolina, Chapel Hill (Other); Indiana University (Other); Medical College of Wisconsin (Other); University of Iowa (Other); Johns Hopkins University (Other); University of Michigan (Other); University of Florida (Other); University of Miami (Other); University of Pennsylvania (Other); Alfred I. duPont Hospital for Children (Other)
Responsible Party: Sponsor
Other Study IDs: 21-018814; RD-2020C22-0338 (Other: PCORI)
Record Dates: First submitted 2021-11-11; First posted 2021-12-27 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Disease Stage 2; Chronic Kidney Disease Stage 3; Pediatric Kidney Disease
Keywords: chronic; child; pediatric; hypertension; proteinuria
MeSH Terms: conditions — Renal Insufficiency, Chronic; Bronchiolitis Obliterans Syndrome; Hypertension; Proteinuria | interventions — Blood Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- angiotensin converting enzyme inhibitors (ACEi) and angiotensin receptor blockers (ARB) categories: The first anti-hypertensive prescribed will be categorized as ACEi, ARB, thiazide diuretic, loop diuretic, beta-blocker, calcium channel blocker, other, and none.
  Interventions: Diagnostic Test: Blood pressure
- Combined renin-angiotensin-aldosterone system (RAAS) blocker category: Secondary analyses will combine ACEi and ARB into a single RAAS blocker category.
  Interventions: Diagnostic Test: Blood pressure
- Urine protein dichotomous indicator: We will determine whether urine protein is evaluated at each encounter and create a dichotomous indicator.
  Interventions: Diagnostic Test: Urine protein

INTERVENTIONS:
Diagnostic Test: Blood pressure — The first anti-hypertensive prescribed will be categorized as ACEi, ARB, thiazide diuretic, loop diuretic, beta-blocker, calcium channel blocker, other, and none; secondary analyses will combine ACEi and ARB into a single RAAS blocker category. We will conduct additional secondary analyses for specific medications with sufficient sample sizes.
  Groups: Combined renin-angiotensin-aldosterone system (RAAS) blocker category; angiotensin converting enzyme inhibitors (ACEi) and angiotensin receptor blockers (ARB) categories
Diagnostic Test: Urine protein — Evaluating urine protein for children with CKD and hypertension is another guideline recommendation, but the frequency, type of assessment (qualitative or quantitative urine protein), and utility for patients without hypertension are unclear. We will determine whether urine protein is evaluated at each encounter and create a dichotomous indicator.
  Groups: Urine protein dichotomous indicator

SUMMARY:
Pediatric chronic kidney disease (CKD) results from health conditions that reduce kidney function for >3 months. It can progress to end-stage kidney disease (ESKD), which requires dialysis or kidney transplant. In adults, CKD is common and caused mainly by hypertension and diabetes. CKD in childhood is rare and caused primarily by congenital anomalies of the genitourinary system and immune-mediated disorders. The best estimate of pediatric CKD prevalence is <1/15,000 pediatric population. Hypertension occurs in 50% of affected children and is a major risk factor for decline in kidney function. Several clinical practice guidelines have offered recommendations for blood pressure (BP) management in pediatric CKD; however, clinical trial and large-scale observational data are limited, leading to a weak evidence base and substantial practice variation. The purpose of PRESERVE is to provide new knowledge to inform shared decision-making regarding BP management for pediatric CKD. We will leverage the Patient-Centered Outcomes Research network (PCORnet®) infrastructure to conduct large-scale observational studies that will address BP management knowledge gaps for pediatric CKD and sub-groups for whom antihypertensive treatment and outcome associations may be different (e.g., cause of kidney disease and proteinuria).

The project's specific aims are:

Aim 1-Enhance the PCORnet Common Data Model (CDM) for pediatric and rare kidney disease research. We will expand and improve the PCORnet CDM with new pediatric- and kidney-specific variables, study-specific data quality optimization, and linkage with the chronic kidney disease in children (CKiD) cohort study and the US Renal Data System (USRDS). CKiD directly measures kidney function [ie, glomerular filtration rate (GFR)] and includes Ambulatory Blood Pressure Monitoring (ABPM). The USRDS provides complete capture of renal replacement therapy [(RRT) dialysis and transplant], two components of the primary clinical outcome.

Aim 2-Describe and examine the effectiveness of consistent BP and urine protein monitoring for preserving kidney function. We will describe the consistency of BP and urine protein monitoring and will contrast clinic BP assessments with ABPM. In longitudinal analyses, we will evaluate the effects of consistent monitoring of BP and urine protein on kidney function decline.

Aim 3-Compare the effectiveness of BP medication strategies for preserving kidney function. We will compare the effects of (1) BP levels when treatment was started, (2) choice of first-line therapies, and (3) ongoing BP control on kidney function decline. We will also assess adverse events related to hypertension management.

Aim 4-Assess patients' lived experiences related to BP management. We will field a survey that examines patient-centered outcomes by level of BP control and medication management approaches. This Aim will provide information on experiences with BP management from the perspectives of patients, parents, and clinicians that will complement the clinical outcomes studied in Aims 2 and 3.

ELIGIBILITY:
Inclusion Criteria:

* Include: patient has an outpatient, ED, or inpatient visit with a physician
* Include: 1 or more eGFR values 30-89 mL/min/1.73m2 using the CKiD U25 formula
* Include: 2 or more eGFR values 30-89 mL/min/1.73m2 on different days using the CKiD U25 formula
* Include: 2 eGFR values in the range 30-89 mL/min/1.73m2 using the CKiD U25 formula greater than or equal to 90 days apart.

Exclusion Criteria:

* Exclude: eGFR value >=90 ml/min using the CKiD U25 formula between the two qualifying eGFRs in mild-moderate range
* Exclude if: Age <1 and >=18 years on CED (see below for definition of CED)
* Exclude if: no nephrologist visit at any time during the study period
* Exclude: if chronic dialysis on or before CED
* Exclude: if kidney transplant on or before CED

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children ages 1 to <18 years with chronic kidney disease stages 2-3 at cohort entrance.
Sampling Method: Non-Probability Sample
Enrollment: 20240 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Decline in estimated glomerular filtration rate (eGFR) | up to 18 months
  Time from cohort entrance (defined as day when first estimated glomerular filtration rate will be measured by the following criteria: (1) >50% decline in eGFR, as measured by the U25 formula; (2) eGFR <=15 ml/min as measured by the U25 formula); (3) initiation of chronic dialysis; or (4) kidney transplant.
  U25 formula: https://doi.org/10.1016/j.kint.2020.10.047

CONTACTS AND LOCATIONS:
Overall Officials: Chris Forrest, MD, Principal Investigator — Children's Hospital of Philadelphia; Michelle Denburg, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Data are from electronic health records, so individual level patient data cannot be shared.